## Data Collection Sheet King Vision Video Laryngoscope aBlade System for Use in Children

| | Patient sticker |
|---|---|
| Subject ID | |
| Date: ASA: I II III | |
| Gender: <b>M F</b> Weight: kg Height: cm | PI or Sub-I: |
| LARYNGEAL VIEW | |
| Cormack Lehane: 1 2 3 4 | |
| INTUBATION | |
| King Vision aBlade size: 1 2 2 channeled Standard laryn | ngoscope blade size: 0 1 2 3 |
| Endotracheal tube size: 2.5 3.0 3.5 4.0 4.5 5.0 5.5 6.0 | Brand: |
| Blade tip position: In valecula Under epiglottis Stylet used: Yes No | |
| Ease of ETT passage: 1 2 3 4 5 (1 = very easy; 2 = easy; 3 = neutral; 4 = difficult; 5 = impossible) | |
| Number of insertion attempts: 1 2 3 (Entry of blade into patient's mouth without the need to remove it once entered) | |
| Insertion time: (Amount of time from Removal of facemask to the first upstroke of etCO <sub>2</sub> ) | |
| Insertion Technique: (check all that apply) [ ] Rotated blade in from side [ ] External laryngeal manipulation [ ] Rotate ETT counterclockwise (channeled only) [ ] Other: | |
| SAE/Complications | |
| Intubation: [ ] Laryngospasm [ ] Gastric Insufflation (Check all that apply) [ ] Bronchospasm [ ] Desaturation (SpO <sub>2</sub> $\leq$ 90%) [ ] Regurgitation/Aspiration [ ] Other: | [ ] None |
| PACU: [ ] Sore throat [ ] Stridor (Check all that apply) [ ] Horseness [ ] Other: [ ] None | |
| Comments: | |

Version: 1.0 Dated: 9-14-15

Signature: